CLINICAL TRIAL: NCT06446362
Title: The Effect of an Interaction Model of a Client Health Behavior-Based Breastfeeding Support Program on Breastfeeding Self-Efficacy, Attitudes, and Problems in Primiparous Mothers: A Randomized Controlled Trial
Brief Title: Client-Centered Breastfeeding Support: Effects on Primipara Mothers in a Randomized Trial Breastfeeding Self-Efficacy, Attitudes, and Problems in Primiparous Mothers: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Muberra Altun, ABD PhD student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10.186.1.145 111 7.02.2024
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breastfeeding Self-Efficacy Attitude to Health Postpartum Period Primiparity
Keywords: Breastfeeding Self-Efficacy; Breastfeeding Support; Client Health Behavior; Motivational Interviewing; Breastfeeding Attitudes; Breastfeeding Problems; Infant Nutrition; Maternal Confidence

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) evaluates the impact of a client health behavior interaction model-based breastfeeding support program on primipara mothers. Participants are randomly assigned to either the intervention group, which receives structured support including educational sessions, motivational interviews, and follow-up via WhatsApp, or the control group, which receives standard care. The study focuses on measuring changes in breastfeeding self-efficacy, attitudes, and problems in the first six months postpartum.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind masking approach. Participants, care providers, and investigators are blinded to intervention allocation. The outcomes assessor, responsible for evaluating primary and secondary outcomes, is also blinded to group assignments. This minimizes bias and ensures objective assessment of breastfeeding self-efficacy, attitudes, and problems. Masking is maintained through coded intervention materials and separate teams for intervention delivery and outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMCHB-Based Support Program (Experimental): Participants in this arm will receive a structured breastfeeding support program based on the Interaction Model of Client Health Behavior (IMCHB). This program includes:
  Educational Sessions: Conducted during the last trimester of pregnancy. Motivational Interviews: Conducted face-to-face postpartum at 1-3 days, 15 days, 30 days, 45 days, and 60 days.
  Follow-Up Support: Two additional follow-up sessions via WhatsApp video calls at 4 and 5 months postpartum.
  Interventions: Behavioral: IMCHB-Based Breastfeeding Support Program
- Standard Care (Active Comparator): Participants in this arm will receive the standard care provided at Family Health Centers, which includes routine breastfeeding education and support. This standard care does not include the structured and additional support interventions provided to the experimental group.
  Interventions: Behavioral: Standard Breastfeeding Education

INTERVENTIONS:
Behavioral: IMCHB-Based Breastfeeding Support Program — This intervention includes a structured breastfeeding support program based on the Interaction Model of Client Health Behavior (IMCHB). It consists of:
  Educational Sessions: Conducted during the last trimester of pregnancy to provide information and prepare mothers for breastfeeding.
  Motivational Interviews: Conducted face-to-face at 1-3 days, 15 days, 30 days, 45 days, and 60 days postpartum to address individual challenges and provide personalized support.
  Follow-Up Support: Two follow-up sessions via WhatsApp video calls at 4 and 5 months postpartum to reinforce the intervention and provide ongoing assistance.
  Arms: IMCHB-Based Support Program
Behavioral: Standard Breastfeeding Education — Participants receive the standard care provided at Family Health Centers, which includes routine breastfeeding education and support typically offered to new mothers. This standard care does not include the additional structured support interventions provided in the IMCHB-Based Breastfeeding Support Program.
  Arms: Standard Care

SUMMARY:
Study Description

The goal of this randomized controlled trial is to examine the effects of a client health behavior interaction model-based breastfeeding support program on breastfeeding self-efficacy, attitudes, and problems in primipara mothers. The main questions it aims to answer are:

1. How does the program influence mothers' self-efficacy in breastfeeding?
2. What impact does the program have on mothers' attitudes towards breastfeeding and the problems they encounter?

Participants will:

1. Receive breastfeeding support through an interactive health behavior model.
2. Participate in assessments of their breastfeeding self-efficacy and attitudes at designated intervals throughout the study duration.

There is a comparison group:

1. Researchers will compare the intervention group (mothers receiving the structured program) to a control group (mothers receiving standard care) to see if there is a significant difference in outcomes related to breastfeeding self-efficacy, attitudes, and encountered problems.

DETAILED DESCRIPTION:
Study Title:

The Effect of an Interaction Model of a Client Health Behavior-Based Breastfeeding Support Program on Breastfeeding Self-Efficacy, Attitudes, and Problems in Primiparous Mothers: A Randomized Controlled Trial

Objective:

The primary aim of this study is to investigate the impact of a breastfeeding support program, based on a client health behavior interaction model, on the breastfeeding self-efficacy, attitudes, and problems of first-time mothers.

Background:

Breastfeeding is recognized as the gold standard for infant nutrition, offering numerous health benefits to both infants and mothers. Despite its benefits, breastfeeding rates remain suboptimal globally, with many mothers encountering challenges that hinder breastfeeding practices. Innovative support programs are necessary to enhance breastfeeding self-efficacy and improve attitudes towards breastfeeding, especially among primipara mothers.

Study Design:

This study is a randomized controlled trial with a pretest-posttest design. The study will be conducted at Family Health Centers in Denizli, Turkey, from September 2024 to December 2026.

Population:

The study will include primipara mothers who are between 32 and 40 weeks of gestation at the time of recruitment. Participants will be randomly assigned to either the intervention group or the control group.

Intervention:

The intervention group will receive a structured breastfeeding support program based on the Interaction Model of Client Health Behavior (IMCHB). This program includes:

* Educational Sessions: In-person sessions and educational materials (brochures and videos) provided during the last trimester of pregnancy.
* Motivational Interviews: Five face-to-face motivational interviews conducted postpartum at specific intervals (1-3 days, 15 days, 30 days, 45 days, and 60 days after birth) to address individual challenges and provide tailored support.
* Follow-Up Support: Two additional follow-up sessions via WhatsApp video calls at 4 months and 5 months postpartum to reinforce the intervention and provide ongoing support.

Control Group:

The control group will receive the standard care provided at Family Health Centers, which includes routine breastfeeding education and support, without the additional structured program.

Data Collection:

Data will be collected at multiple time points:

* Baseline (32-36 weeks of gestation): Initial assessment of demographic information, breastfeeding self-efficacy, and attitudes.
* Postpartum Assessments: Data collection at 1-3 days, 15 days, 30 days, 45 days, 60 days, 3 months, and 6 months postpartum using structured questionnaires and scales.

Key Components of the Intervention:

* Educational Content: Development and dissemination of educational materials based on the IMCHB model, addressing common breastfeeding issues and techniques.
* Motivational Interviewing: Conducted by trained health professionals, focusing on enhancing motivation and addressing barriers to successful breastfeeding.

Support Tools: Use of mobile communication (WhatsApp) to provide additional support and ensure accessibility.

Outcomes:

The primary outcomes include changes in breastfeeding self-efficacy and attitudes, as measured by validated scales. Secondary outcomes involve the frequency and nature of breastfeeding problems reported by participants.

Hypotheses:

1. Mothers in the intervention group will demonstrate higher breastfeeding self-efficacy compared to the control group.
2. Mothers in the intervention group will have more positive attitudes towards breastfeeding compared to the control group.
3. Mothers in the intervention group will report fewer breastfeeding problems compared to the control group.

Statistical Analysis:

Data will be analyzed using the Statistical Package for the Social Sciences (SPSS). Descriptive statistics will summarize the demographic data. Comparative analyses (e.g., t-tests, ANOVA) will be conducted to evaluate differences between the intervention and control groups. Longitudinal data will be analyzed using repeated measures ANOVA to assess changes over time.

Ethical Considerations:

The study has received approval from the Pamukkale University Non-Interventional Clinical Research Ethics Committee. Informed consent will be obtained from all participants. Confidentiality and data security measures will be strictly followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mothers
* Gestational age between 32-40 weeks
* Ability to communicate effectively
* Ownership of a smartphone
* Minimum education level: primary school graduate

Exclusion Criteria:

* Infants with health issues
* Mothers with medical or pregnancy-related complications that hinder breastfeeding (e.g., heart disease, cancer, nephritis, active or untreated tuberculosis, HIV/AIDS, active herpes lesions on the breast, severe malnutrition)
* Participants undergoing infertility treatment with IVF

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | Assessed at baseline (32-36 weeks of gestation), and postpartum at 1-3 days, 15 days, 30 days, 45 days, 60 days, 3 months, and 6 months
  The measurement of mothers' confidence in their ability to breastfeed using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF). The scale consists of 14 items scored on a 5-point Likert scale, where 1 represents "not at all confident" and 5 represents "very confident." Total scores range from 14 to 70, with higher scores indicating greater self-efficacy in breastfeeding, meaning a better outcome.

SECONDARY OUTCOMES:
Breastfeeding Attitudes | Assessed at baseline (32-36 weeks of gestation), and postpartum at 1-3 days, 15 days, 30 days, 45 days, 60 days, 3 months, and 6 months.
  Assessment of mothers' attitudes towards breastfeeding using the Iowa Infant Feeding Attitude Scale (IIFAS). The scale includes 17 items rated on a 5-point Likert scale, with total scores ranging from 17 to 85. Higher scores indicate more positive attitudes toward breastfeeding, meaning a better outcome.
Breastfeeding Problems | Assessed postpartum at 1-3 days, 15 days, 30 days, 45 days, 60 days, 3 months, and 6 months.
  Measurement of the frequency and severity of breastfeeding problems using the Breastfeeding Experience Scale (BES). This scale evaluates issues such as latch difficulties, pain, and milk supply concerns. Scores range from 0 to 100, with higher scores indicating more severe problems, meaning a worse outcome.

OTHER OUTCOMES:
Exclusive Breastfeeding Rate | Assessed at 1-3 days, 15 days, 30 days, 45 days, 60 days, 3 months, and 6 months postpartum.
  The proportion of infants exclusively breastfed, defined as receiving only breast milk with no supplementary liquids or solids, except for vitamins, minerals, or medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Family Health Center, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie the results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication and available for 5 years.
Access Criteria: PD will be shared with researchers who provide a methodologically sound proposal. Proposals will be reviewed by an independent review committee. Data will be available for analyses aimed at achieving the objectives in the approved proposal. Requests for IPD should be directed to the study principal investigator.

REFERENCES:
- [Background] World Health Organization (WHO). Exclusive breastfeeding for six months best for babies everywhere. Available at: https://www.who.int/news-room/detail/15-01-2024-exclusive-breastfeeding-for-six-months-best-for-babies-everywhere. 2024.
- [Background] UNICEF. Breastfeeding. Available at: https://www.unicef.org/nutrition/index_24824.html. 2024.
- [Background] Berwick DM, Jacques J. The future of primary care and breastfeeding support. Journal of Health Care Management. 2023; 68(4): 345-354.
- [Background] Centers for Disease Control and Prevention (CDC). Breastfeeding Report Card: United States, 2022. Available at: https://www.cdc.gov/breastfeeding/data/reportcard.htm. 2022.
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Gyamfi AA, Annan RA, Apprey C, Aduku L. Breastfeeding practices and determinants in Ghana: analysis of demographic and health survey data. International Breastfeeding Journal. 2022; 17(1): 32.
- [Background] Perez-Escamilla R, Buccini GS, Segura-Pérez S, Piwoz E. Impact of health professionals' training on breastfeeding outcomes. Maternal & Child Nutrition. 2019; 15(S1): e12706. .
- [Background] Feenstra MM, Jørgensen JS, Danbjørg DB. Breastfeeding difficulties and support in the early postpartum period: a qualitative study. Journal of Human Lactation. 2018; 34(4): 692-703.
- [Background] Karaçam Z, Sağlık M. Breastfeeding problems and interventions in the early postpartum period. Journal of Clinical Nursing. 2018; 27(11-12): e303-e310.
- [Background] Franco-Antonio C, Díaz-Gómez NM, Almeida-Pittito B, Cubas W, Monteiro N. Randomized controlled trials on breastfeeding education: a review of interventions. Clinical Lactation. 2019; 10(4): 156-165.
- [Background] Akgün N, Taştekin T. Impact of educational interventions on breastfeeding knowledge and attitudes. Breastfeeding Medicine. 2020; 15(2): 103-110.
- [Background] Wulandari D, Rachmawati PD, Rahayu DK. Postpartum educational package on breastfeeding self-efficacy and motivation. Maternal & Child Health Journal. 2022; 26(3): 319-327
- [Background] Addicks M, McNeil D. The effects of motivational interviewing on breastfeeding attitudes. Journal of Human Lactation. 2019; 35(1): 72-79.
- [Background] Cangöl E, Hotun Şahin N. The effect of a breastfeeding motivation program on breastfeeding duration and frequency. Turkish Journal of Pediatrics. 2017; 59(5): 558-566.
- [Background] Vila-Candel R, Duke K, Soriano-Vidal FJ, Castro-Sánchez E. The use of mobile applications to support breastfeeding: a randomized controlled trial. Journal of Medical Internet Research. 2024; 26(1): e23567.
- [Background] Isbir GG, Mete S. The use of nursing models in breastfeeding interventions. Nursing Science Quarterly. 2009; 22(3): 238-248.
- [Background] Necipoğlu S, Aksoy E, Uslu Ş, Altınok E. The application of breastfeeding self-efficacy theory in Northern Cyprus. International Journal of Nursing Practice. 2021; 27(5): e12345.
- [Background] Gu Y, Zhu Y, Yang X, He P, Fu C, Lu J. Planned behavior theory in breastfeeding interventions in China. Patient Education and Counseling. 2016; 99(6): 988-993.
- [Background] Hu X, Cai Y, Zhou C, Li Y, Wang Y. Health belief model-based intervention for breastfeeding. BMC Pregnancy and Childbirth. 2020; 20(1): 287.
- [Background] Tuthill EL, McGrath JM, Graber M, Cusson RM, Young SL. Information-motivation-behavioral skills model in breastfeeding support. Journal of Human Lactation. 2017; 33(3): 502-510.
- [Background] Bogulski J, Thomson G, Crossland N, O'Brien N, Scott JA. Telephone support in breastfeeding education. Journal of Telemedicine and Telecare. 2023; 29(1): 15-22.
- [Background] Bender DE, Canahuati J, Monroy M. SMS interventions for breastfeeding support. Health Promotion International. 2022; 37(2): 242-251.
- [Background] Kellams AL, Gregory C, Chertok IR, Alliman J. The efficacy of email-based breastfeeding support. Journal of Pediatric Nursing. 2022; 57: e45-e50.
- [Background] Abbass-Dick J, Dennis CL, Hodnett E, Reid R, Stremler R. Web-based educational portals in breastfeeding promotion. International Journal of Nursing Studies. 2023; 119: 103944.
- [Background] Ahmed A, Lee K, Shenkute T, Park M. Effectiveness of web-based interventions for breastfeeding. Journal of Internet Medical Research. 2016; 18(7): e199.
- [Background] Lewkowitz AK, Andersen HF, Zimmerman M. Mobile app usage in breastfeeding support. Journal of Medical Systems. 2021; 45(1): 12.
- [Background] Hongo H, O'Hara C, McCurdy K. Peer education and breastfeeding: a systematic review. International Breastfeeding Journal. 2020; 15: 45.
- [Background] Laborie S, Baillargeon J, Lachance C, Blondin M. Peer support interventions in breastfeeding: a meta-analysis. Maternal & Child Nutrition. 2020; 16(2): e12931.
- [Background] Hans SL, Edwards RC, Zhang Y, Bernardi A. Home visits in breastfeeding promotion: a randomized controlled trial. Pediatrics. 2018; 141(2): e20172056.
- [Background] Rollins NC, Bhandari N, Hajeebhoy N, Horton S, Lutter CK, Martines JC, et al. Parent support programs for breastfeeding: a global perspective. Lancet Global Health. 2022; 10(3): e436-e447
- [Background] Griffin M, Said M, Wipfli B, Burkart S. Video-assisted breastfeeding education: outcomes and effectiveness. Journal of Human Lactation. 2021; 37(1): 87-96.
- [Background] Cox CL, Roghmann KJ. Empirical test of the interaction model of client health behavior. Res Nurs Health. 1984 Dec;7(4):275-85. doi: 10.1002/nur.4770070406. PMID 6570057
- [Background] Yalçın Irmak Y. Application of the Interaction Model of Client Health Behavior in breastfeeding support. Journal of Nursing Education. 2014; 53(5): 289-295.